CLINICAL TRIAL: NCT00889460
Title: Phase I Study to re-Investigate the Safety, Tolerability and Pharmacodynamic Effects of SLIT(Tablets) With Recombinant Bet v1 Given in Single Rising Doses and in Multi Dose Regimens to Subjects Sensitised to Birch Pollen
Brief Title: Safety and Tolerability Study of rBet v1 SLIT Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stallergenes Greer (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Bruno ROBIN, Stallergenes S.A.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VO58.07 DK
Record Dates: First submitted 2009-04-28; First posted 2009-04-29 (Estimated); Last update posted 2009-04-29 (Estimated); Status verified 2009-04

CONDITIONS: Birch Pollen-Related Rhinoconjunctivitis; Rhinitis, Allergic, Seasonal
Keywords: rBet v 1; Birch pollen allergy; Sublingual Immunotherapy
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Placebo group
  Interventions: Biological: Placebo
- 2 (Experimental): rBet v 1 tablets
  Interventions: Biological: rBet v 1

INTERVENTIONS:
Biological: rBet v 1 — Two tablets (1 placebo + 1 rBet v 1 or 2 rBet v 1) were administered every day over 2 weeks with a 2-day break for the week-end. Administered doses ranged from 12.5 to 100 µg rBet v 1.
  Other Names: rBet v 1.0101
  Arms: 2
Biological: Placebo — Two matching placebo tablets were administered every day over 2 weeks with a 2-day break for the week-end.
  Arms: 1

SUMMARY:
The purpose of this study is to determine the safety and tolerability of several doses of r Bet v1 administered as sub-lingual tablets in subjects sensitised to birch pollen.

ELIGIBILITY:
Inclusion Criteria:

* written consent
* Male or female subject from 18 to 60 years old and in general good health
* For woman of child bearing potential:
* Symptoms of birch pollen induced allergic rhinitis for at least the last 2 years.
* Sensitisation to birch pollen as demonstrated with a positive SPT to birch pollen and specific IgE level (birch pollen and r Bet v1) >0.70 kU/L at screening.
* FEV1 at least of 80% of predicted values at screening.
* Subject accepting to comply fully with the protocol.

Exclusion Criteria:

* Past or current disease which as judged by the Investigator, may affect the outcome of this study.
* History of life-threatening asthma,
* Asthma requiring daily treatment (whatever the pharmaceutical class).
* Pregnant or lactating woman.
* Subject being treated with inhaled steroids within 4 weeks prior to screening visit or within 12 weeks prior to screening visit.
* Subject who previously received desensitisation treatment to birch pollen and/or other betulaceae (e.g., hazel tree, alder) or who plan to start desensitisation treatment during this study.
* Symptoms during the treatment phase due to a sensitivity to a second allergen.
* Subjects treated with ongoing immunotherapy with another allergen

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2007-11; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Local tolerability | Assessed every day over 2 weeks
Global safety | Assessed every day over 2 weeks

SECONDARY OUTCOMES:
Immunological markers (IgE and IgG4) | Between selection and follow-up visit (up to 18 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Jorgen MALLING, Pr. MD, Principal Investigator — National University Hospital - Copenhagen - DENMARK
Locations (1):
- National University Hospital - Allergy Unit 4222, Copenhagen, Denmark

REFERENCES:
- [Result] L. Winther, L.K. Poulsen, B. Robin, M. Mélac, H. Malling Safety and Tolerability of Recombinant Bet v 1 (rBet v 1) Tablets in Sublingual Immunotherapy (SLIT) The Journal of Allergy and Clinical Immunology February 2009 (Vol. 123, Issue 2, Page S215)